CLINICAL TRIAL: NCT03084419
Title: Safety of Abatacept in Rheumatoid Arthritis Associated Interstitial Lung Disease: A Feasibility Trial
Brief Title: APRIL (AbatacePt in Rheumatoid Arthritis-ILD)
Acronym: APRIL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Frances Hall, Consultant Rheumatologistand and Clinical Lead for Connective Tissue Disease, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APRIL
Record Dates: First submitted 2017-03-07; First posted 2017-03-21 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease
Keywords: Rheumatoid Arthritis; Interstitial Lung Disease; RA-ILD; Abatacept
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: The investigators will perform a small clinical trial to assess the feasibility of performing a larger randomised controlled trial.
  Thirty participants with RA-ILD will be treated with abatacept infusions, which will be given fortnightly for the first 4 weeks, then every 4 weeks for a total of 20 weeks.
  Participants will sign informed consent at visit 1 (screening visit). There is then a 28 day window before treatment starts at visit 2 (baseline). Each participants participation in the trial is estimated to last 28 weeks from visit 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abatacept in patients with RA-ILD (Experimental): Thirty participants with RA-ILD will be treated with abatacept infusions, which will be given fortnightly for the first 4 weeks, then every 4 weeks for a total of 20 weeks.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — The IV dose varies according to weight:
  <60kg=500mg
  ≥60 but≤100kg=750mg >100kg=1g
  This equates to approximately 10mg/kg.
  Other Names: Orencia

SUMMARY:
Early initiation of treatment for Rheumatoid arthritis (RA) can prevent several of the long term problems associated with the condition. However, many RA patients develop lung inflammation and scarring, called 'interstitial lung disease' (RA-ILD), contributing to early death in 1 in 5 people. There is no proven treatment for these patients and some medications for RA can in fact worsen their lung disease. There is a need therefore to find safe medications that can not only control RA joint disease, but also prevent progression of RA-ILD. Abatacept is an approved drug for treating RA and is used widely. It is a newer RA medication, with a unique mechanism of action, and it has been shown to prevent progression of joint damage and improve physical function. The investigators aim to assess the safety of this medication in patients with RA-ILD and improve our understanding of the mechanism of lung damage in rheumatoid disease.

The investigators will perform a small clinical trial to assess the feasibility of performing a larger randomized controlled trial. A total of 30 patients with RA-ILD will be treated with abatacept infusions fortnightly for the first month, then every 4 weeks for a total of 20 weeks. In order to be eligible for the study, a patient must be able to provide written informed consent, be aged ≥18 years, and have interstitial lung disease that has not responded to or progressed over 6 months despite conventional immunosuppression. Change in lung function (forced vital capacity) at 24 weeks will be evaluated. To assess the mechanisms that may be involved with the development of ILD, the investigators will assess the effects of abatacept on biomarkers obtained from the blood and the lung (bronchoalveolar lavage), including markers of infection (the lung microbiome).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Agree to use 2 acceptable forms of effective contraception for the duration of the study trial and a further 14 weeks after completion
* Meet a diagnosis of RA by 2010 EULAR/ACR criteria
* Have interstitial lung disease associated with RA, with supportive findings on their PFTs and CT Chest scans. Participants will be included if their ILD has progressed over 14 months. Progression will be defined as EITHER:
* A decrease in FVC by at least 5% when comparing two sets of PFTs done in the last 24 months, but with an interval of up to 14 months between the PFTs OR
* Progression of lung fibrosis on a high-resolution CT chest, as reported by a chest radiologist.

Exclusion Criteria:

* Unable to provide informed written consent
* Participants who are taking other immunosuppressants, e.g. mycophenolate mofetil (MMF), unless this has been discontinued with an adequate washout period. The exceptions to this exclusion criterion are methotrexate (MTX) and hydroxychloroquine, which are allowed provided the dose has been stable for 6 weeks prior to baseline (visit 2).
* Participants who have been taking > 10mg Prednisolone daily within the last 6 weeks prior to baseline (visit 2)
* Participants who have had rituximab, within the 24 weeks prior to baseline (Visit 2)
* Any participant with active signs or symptoms of infection at the baseline (visit 2) or requiring antibiotic treatment within the preceding 4 weeks
* Any participant with significant co-existing lung disease, such as asthma, bronchiectasis, emphysema, Chronic Obstructive Pulmonary Disease (COPD) or if their pre-bronchodilator FEV1/FVC ratio is < 60%.
* Significant other co-morbidity (e.g. active malignancy/liver disease/renal disease) within the last 5 years
* Prior use of abatacept at any time
* Participation in any other clinical trial within 8 weeks or 5 half-lives of IMP, whichever is longer, prior to baseline (visit 2) (participation in 'observational' studies is allowed)
* Hypersensitivity to any excipients of abatacept
* Any participant who has had live vaccines within 6 weeks prior to baseline (Visit 2)
* Participant is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 28 weeks (Screening-V9)
  Assessing the change of Forced Vital Capacity (FVC) across screening, baseline V2 (prior to abatacept), V6 and V9.

SECONDARY OUTCOMES:
Transfer factor of the lung for carbon monoxide (TLCO) | 28 weeks (Screening-V9)
  Assessing the change of Transfer factor of the lung for carbon monoxide (TLCO) at screening (prior to abatacept), V6 and V9.
MRC dyspnoea score | 24 weeks (Baseline-V9)
  Assessing the change of MRC dyspnoea score completed at Baseline V2 (prior to abatacept), V6, V9
Kings Brief Interstitial Lung Disease score (K-BILD) | 24 weeks (Baseline-V9)
  Assessing the change of Kings Brief Interstitial Lung Disease score (K-BILD) questionnaire completed at Baseline V2 (prior to abatacept), V6, V9
Semi-quantitative radiological scoring of the ILD | 28 weeks (Screening-V9)
  Assessing the change of HRCT chest scans performed at screening (prior to abatacept and V9 (end of trial)
Resting oxygen saturation | 28 weeks
  Resting oxygen saturation recorded at all visits
DAS28 | 28 weeks
  DAS28 recorded at all visits
Leicester Cough Questionnaire score | 24 weeks (Baseline-V9)
  Assessing the change of Leicester Cough Questionnaire completed at Baseline V2 (prior to abatacept), V6, V9
EQ-5D | 24 weeks (Baseline-V9)
  Assessing the change of EQ-5D Questionnaire completed at Baseline V2 (prior to abatacept), V6, V9
Respiratory tract infection | 24 weeks (Baseline-V9)
  Assessing the number of Respiratory tract infections recorded following IMP dosing between V2-V9

CONTACTS AND LOCATIONS:
Overall Officials: Frances Hall, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Addenbrookes Hospital, Cambridge
  - Papworth Hospital, Cambridge

IPD SHARING:
Plan to Share IPD: No